CLINICAL TRIAL: NCT00740246
Title: A Multi-Center, Randomized, Blinded, Placebo Controlled, Cross-Over Study to Investigate the Safety and Tolerability of Intravenous VIT-45 in Patients With Iron Deficiency Anemia
Brief Title: Safety and Tolerability of Intravenous VIT-45 in Patients With Iron Deficiency Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1VIT05006
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VIT-45 on Day 0, then Placebo on Day 7 (Experimental): Day 0: 15 mg/kg up to a maximum dose of 1,000 mg of iron as VIT-45 over 15 minutes intravenously.
  Day 7: for weight >33 kg, 250 cc of normal saline and for weight ≤33 kg, 100 cc of normal saline over 15 minutes intravenously.
  Interventions: Drug: VIT-45; Drug: Placebo
- Placebo on Day 0, then VIT-45 on Day 7 (Experimental): Day 0: for weight >33 kg, 250 cc of normal saline and for weight ≤33 kg, 100 cc of normal saline over 15 minutes intravenously.
  Day 7: 15 mg/kg up to a maximum dose of 1,000 mg of iron as VIT-45 over 15 minutes intravenously.
  Interventions: Drug: VIT-45; Drug: Placebo

INTERVENTIONS:
Drug: VIT-45 — 15 mg/kg up to a maximum dose of 1,000 mg of iron as VIT-45 over 15 minutes intravenously
  Other Names: ferric carboxymaltose
Drug: Placebo — for weight >33 kg, 250 cc of normal saline and for weight ≤33 kg, 100 cc of normal saline over 15 minutes intravenously

SUMMARY:
The objective of this study is to evaluate the safety and tolerability of VIT-45 in the treatment of Iron Deficiency Anemia

DETAILED DESCRIPTION:
Evaluate the safety and tolerability of VIT-45 in the treatment of Iron Deficiency Anemia

ELIGIBILITY:
Inclusion Criteria:

* Subjects > or = 18 years of age and able to give informed consent
* Historical laboratory Hgb indicative of anemia within 3 months prior to screening visit
* Screening Visit laboratory Hgb indicative of anemia
* Screening Visit ferritin indicative of iron deficiency anemia

Exclusion Criteria:

* Known hypersensitivity to VIT-45
* Previously received VIT-45
* Parenteral iron in the 4 weeks prior to screening
* Chronic or serious active infection
* Malignancy history
* Aspartate aminotransferase (AST) or Alanine transaminase( ALT) greater than the upper limit of normal
* Anticipated need for surgery or initiation of dialysis during the study
* Pregnant or sexually active females who are not willing to use an effective form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2005-07 (Actual); Primary Completion 2006-02 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bregman, MD, Study Director — American Regent, Inc.
Locations (1):
- Luitpold Pharmaceuticals, Norristown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Seid MH, Valaoras TG, Barish CF, Dinh Q. Safety Profile of Ferric Carboxymaltose, a New High Dose Intravenous Iron in Patients with Iron Deficiency Anemia. Society for the Advancement of Blood Management 2007.
- [Result] Seid MH, Mangione A, Valaoras TG, Anthony LB, Barish CF. Safety Profile of Ferric Carboxymaltose, a New High Dose Intravenous Iron in Patients with Iron Deficiency Anemia. Society for the Advancement of Blood Management 2007.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and medical clinics
Groups:
- VIT-45/Placebo: VIT-45 (15 mg/kg up to a maximum of 1000 mg) given on Day 0. After a washout period of 1 week, they then received Placebo on Day 7
- Placebo/VIT-045: Placebo given on Day 0. After a washout period of 1 week, they then received VIT-45 (15 mg/kg up to a maximum of 1000 mg) given on Day 0.
Period: Overall Study
Arm/Group | VIT-45/Placebo | Placebo/VIT-045
Started | 305 | 289
Completed | 291 | 277
Not Completed | 14 | 12
Not completed — Received Blood Transfusion | 0 | 1
Not completed — Adverse Event | 1 | 2
Not completed — Selection Criteria/Study Compliance | 2 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Withdrawn By Site Due To non-compliance | 1 | 0
Not completed — Discontinued Due To Hurricane Related Issue | 1 | 1
Not completed — Unable To Perform Venipuncture For Day 7, Day 14 Labs, and Day 7 Infusion | 1 | 0
Not completed — Unable To Comply With Study Visits | 2 | 0
Not completed — Unable to Access Vein | 0 | 2
Not completed — Early Term - Patient could not return for second infusion due to Thanksgiving Holiday | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: All subjects who received at least 1 dose of randomized study drug
Groups:
- VIT-45: VIT-45 given on Day 0 and Placebo on Day 7. For assessment purposes, this arm included all subjects who received VIT-45 at Day 0 and Day 7. Also included in this assessment was 12 pharmacokinetic (PK) patients. The PK portion of the study was open-label, not part of the cross-over design, where subjects received 1 unblinded dose of VIT-45 at Day 0. Select sites participated and subjects were enrolled if they agreed to the extra blood draws.
- Placebo: Placebo given on Day 0 and VIT-45 on Day 7. For assessment purposes, this arm included all subjects who received Placebo at Day 0 and Day 7.
- Total: Total of all reporting groups
Arm/Group | VIT-45 | Placebo | Total
Number analyzed (Participants) | 305 | 289 | 594
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (16.4325) | 42.6 (16.9296) | 41.9 (16.6767)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 70
  Male | 269 | 255 | 524
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 49 | 52 | 101
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 190 | 178 | 368
  White | 62 | 48 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 11 | 15
Region of Enrollment [Number; unit: participants]
  United States | 305 | 289 | 594
Weight [Mean (Standard Deviation); unit: kilograms] | 80.6 (80.6) | 80.6 (80.6) | 80.6 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events During Each 7-day Study Period
Description: Number of participants with any treatment-emergent adverse events experienced by participants. The 7-day study period for Study Period 1 ended with the initiation of dosing for Study Period 2. The 7-day study period fo Study Period 2 ended with the completion of Day 14 procedures.
Time Frame: Day 0 to 7
Population: At Least 1 Treatment-Emergent Adverse Event
Measure: Number; unit: participants
Groups:
- ViT-45: VIT-45 given on Day 0 or Day 7
- Placebo: Placebo given on Day 0 or Day 7.
Arm/Group | ViT-45 | Placebo
Number analyzed (Participants) | 584 | 569
participants | 174 | 114

ADVERSE EVENTS:
Time Frame: 7 days
Description: 594 who received at least 1 dose of study medication were included in the Safety Population (SP). For VIT-45 exposure, 10 subjects that were scheduled to receive VIT-45 as a 2nd dose did not (582-10 = 572 safety exposures from crossover portion). After including the 12 PK subjects, a total of 584 subjects were included in the SP. For the placebo exposure, 13 subjects that were scheduled to receive placebo as a 2nd dose did not did not (582-13 = 569 safety exposures from crossover portion).
Groups:
- VIT-45 on Day 0 or Day 7: Participants received VIT-45 on either Day 0 or Day 7 (a maximum dose of 1,000 mg of iron as VIT-45 over 15 minutes intravenously)
- Placebo on Day 0 or Day 7: Participants received Placebo on Day 0 or Day 7 (for weight >33 kg, 250 cc of normal saline and for weight ≤33 kg, 100 cc of normal saline over 15 minutes intravenously)
Arm/Group | VIT-45 on Day 0 or Day 7 | Placebo on Day 0 or Day 7
All-Cause Mortality (participants affected / at risk) | 1/584 | 0/569
Serious Adverse Events (participants affected / at risk) | 2/584 | 4/569
Other Adverse Events (participants affected / at risk) | 31/584 | 19/569
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VIT-45 on Day 0 or Day 7 (N=584) | Placebo on Day 0 or Day 7 (N=569)
Pneumonia (Infections and infestations) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Diabetes mellitus non-insulin dependent (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Endometritis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VIT-45 on Day 0 or Day 7 (N=584) | Placebo on Day 0 or Day 7 (N=569)
Headache (Nervous system disorders) | 31 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less